CLINICAL TRIAL: NCT05783596
Title: A Phase 2 Study of Glofitamab and Obinutuzumab for First-line Treatment of Follicular Lymphoma and Marginal Zone Lymphoma
Brief Title: Glofit and Obin in Follicular Lymphoma and Marginal Zone Lymphoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Reid Merryman, MD (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Reid Merryman, MD, Principal Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-632
Record Dates: First submitted 2023-03-13; First posted 2023-03-24 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Follicular Lymphoma; Marginal Zone Lymphoma; Indolent Non-hodgkin Lymphoma
Keywords: Follicular Lymphoma; Marginal Zone Lymphoma; Indolent Non-hodgkin Lymphoma; Immunotherapy
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone | interventions — obinutuzumab; glofitamab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Obinutuzumab + Glofitamab for Follicular Lymphoma (Experimental): Participants will undergo study procedures as outlined:
  * Imaging scans (CT or PET) at screening and after cycles 3, 7, and 12 of treatment.
  * Bone marrow biopsy at baseline.
  * Cycle 1
    * Days -21, -14, -7, 0 of 36 day cycle: Predetermined dose of Obinutuzumab.
    * Days 1 and 8 of 36 day cycle: Predetermined dose of Glofitamab. (First dose will be administered in the hospital.)
  * Cycles 2 - 12:
    o Day 1 of 21 day cycle: Predetermined dose of Glofitamab.
  * Bone marrow biopsy within 2 weeks of end of treatment.
  * Imaging scans (CT or PET) at 12, 18, and 24 months after treatment initiation.
  * Follow up visits up to 5 years after treatment completion.
  Interventions: Drug: Obinutuzumab; Drug: Glofitamab
- Obinutuzumab + Glofitamab for Marginal Zone Lymphoma (Experimental): Participants will undergo study procedures as outlined:
  * Imaging scans (CT or PET) at screening and after cycles 3, 7, and 12 of treatment.
  * Bone marrow biopsy at baseline.
  * Cycle 1
    * Days -21, -14, -7, 0 of 36 day cycle: Predetermined dose of Obinutuzumab.
    * Days 1 and 8 of 36 day cycle: Predetermined dose of Glofitamab. (First dose will be administered in the hospital.)
  * Cycles 2 - 12:
    o Day 1 of 21 day cycle: Predetermined dose of Glofitamab.
  * Bone marrow biopsy within 2 weeks of end of treatment.
  * Imaging scans (CT or PET) at 12, 18, and 24 months after treatment initiation.
  * Follow up visits up to 5 years after treatment completion.
  Interventions: Drug: Obinutuzumab; Drug: Glofitamab

INTERVENTIONS:
Drug: Obinutuzumab — Humanized glycoengineered type II anti-CD20 monoclonal antibody, via IV infusion.
  Other Names: RO5072759, GA101, GAZYVA, GAZYVARO
Drug: Glofitamab — T-cell bispecific humanized monoclonal antibody, via IV infusion.
  Other Names: RO7082859

SUMMARY:
The purpose of this study is to determine how effective and safe the combination of glofitamab and obinutuzumab is in treating patients with Follicular Lymphoma (FL) and Marginal Zone Lymphoma (MZL) who have not received other treatments for their lymphoma.

The names of the study drugs involved in this study are:

* Glofitamab (a type of immunotherapy)
* Obinutuzumab (a type of immunotherapy)

DETAILED DESCRIPTION:
This is an open-label, multicenter, phase II study to evaluate the efficacy and safety of obinutuzumab and glofitamab for patients with untreated follicular lymphoma (FL) or marginal zone lymphoma (MZL). Obinutuzumab and Glofitamab use the immune system to target and attack cancer cells.

The research study procedures include screening for eligibility, study treatment visits, bone marrow biopsies, blood tests, Computerized Tomography (CT) scans, and Positron Emission Tomography (PET) scans.

The U.S. Food and Drug Administration (FDA) has not approved glofitamab as a treatment for any disease.

The U.S. FDA has approved obinutuzumab in combination with chemotherapy for patients with follicular lymphoma.

Participants will receive study treatment for approximately 9 months and will be followed for 10 years.

It is expected that about 45-50 people will take part in this research study.

Genentech and Roche are supporting this research study by providing the study drugs, glofitamab and obinutuzumab, and funding for the study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of either FL (grade 1-3A) or MZL (any subtype) with review of the diagnostic pathology specimen at one of the participating institutions. Patients with active histologic transformation are excluded.
* No prior systemic therapy for FL or MZL. Prior treatment with radiation therapy or short course steroids is allowed.
* Meets at least one criterion to begin treatment based on the modified GELF criteria:

  * Symptomatic adenopathy
  * Organ function impairment due to disease involvement, including cytopenias due to marrow involvement (WBC <1.5x109/L; absolute neutrophil count [ANC] <1.0x109/L, Hgb <10g/dL; or platelets <100x109/L)
  * Constitutional symptoms
  * Maximum diameter of disease > 7cm
  * >3 nodal sites of involvement
  * Risk of local compressive symptoms
  * Splenomegaly (craniocaudal diameter > 16cm on CT imaging)
  * Clinically significant pleural or peritoneal effusion
  * Leukemic phase (>5x109/L circulating malignant cells)
  * Rapid generalized disease progression
  * Renal infiltration
  * Bone lesions
* Patients cannot be in need of urgent cytoreductive chemotherapy in the opinion of the treating investigator.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2. (Appendix A)
* Age ≥18 years.
* Adequate hematologic and organ function:

  * Absolute neutrophil count > 1.0x109/L unless due to marrow involvement by lymphoma in which case ANC must be >0.5x109/L
  * Platelets > 75 x109/L, unless due to marrow involvement by lymphoma, in which case platelets must be >50 x109/L
  * Creatinine clearance > 40ml/min (by Cockcroft-Gault Formula)
  * Total bilirubin < 1.5 X ULN, unless Gilbert syndrome, in which case direct bilirubin must be < 1.5 x ULN
  * AST/ALT < 2.5 X ULN, unless documented liver involvement by lymphoma, in which case AST/ALT must be <5 x ULN
* Ability to understand and the willingness to sign a written informed consent document.
* Willingness to provide a pre-treatment tumor sample by core needle or excisional surgical biopsy. A fresh biopsy is strongly encouraged, but an archival sample is acceptable if the following provisions are met: 1) availability of a tumor-containing formalin-fixed, paraffin-embedded (FFPE) tissue block, 2) if the tumor containing FFPE tissue block cannot be provided in total, sections from this block should be provided that are freshly cut and mounted on positively-charged glass slides (SuperFrost Plus are recommended). Preferably, 25 slides should be provided; if not possible, a minimum of 15 slides is required. Exceptions to this criterion may be made with approval of the sponsor-investigator.
* Willingness to remain abstinent or to use two effective contraceptive methods that result in a failure rate of <1% per year from screening until: (a) at least 3 months after pre-treatment with obinutuzumab or 2 months after the last dose of glofitamab, whichever is longer, if the patient is a male or (b) until at least 18 months after pre-treatment with obinutuzumab or 2 months after the last dose of glofitamab, whichever is longer, if patient is a female. Examples of contraceptive methods with a failure rate of <1% per year include:

  * Tubal ligation, male sterilization, hormonal implants, established proper use of hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices.
  * Alternatively, two methods (e.g., two barrier methods such as a condom and a cervical cap) may be combined to achieve a failure rate of <1% per year. Barrier methods must always be supplemented with the use of a spermicide.

Exclusion Criteria:

* Patients who require systemic immunosuppressive therapy for an ongoing medical condition will be excluded. For corticosteroids, patients receiving a prednisone dose of >10 mg daily (or equivalent) will not be eligible. A short course of steroids (up to 14 days, not exceeding 40 mg dexamethasone or equivalent in a single day) for symptom palliation is allowed, in which case patients should be off steroids at least 7 days prior to treatment start.
* Patients with bulky cervical adenopathy that is 1) compressing the upper airway or 2) in close proximity to the upper airway and could result in airway compression during a tumor flare event).
* History of severe allergic or anaphylactic reactions to monoclonal antibody therapy unless in consultation with an allergy specialist they are deemed eligible for retreatment with desensitization.
* Patients, who have had a major surgery or significant traumatic injury within 4 weeks of start of study drug, patients who have not recovered from the side effects of any major surgery (defined as requiring general anesthesia).
* Patients with known HIV infection or hepatitis B or C infection. Testing for HIV is optional. Testing for hepatitis B and C is mandatory. Patients with hepatitis B core Ab positivity but negative surface antigen and negative viral load may be enrolled if they can be treated with a prophylactic agent (e.g., entecavir); patients with hepatitis C seropositivity who have a negative viral load can also be enrolled.
* Patients with a systemic fungal, bacterial, viral, or other infection not controlled (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment).
* Prior history of another malignancy (except for non-melanoma skin cancer or in situ cervical or breast cancer) unless disease free for at least 2 years. Patients with prostate cancer (Gleason score 6-7) are allowed if PSA is less than 1 ng/mL.
* Patients should not have received immunization with lives or live attenuated vaccine within one week of study entry or during study period.
* Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study or limit adherence to study requirements.
* Patients with any one of the following currently on or in the previous 6 months will be excluded: myocardial infarction, congenital long QT syndrome, torsade de pointes, unstable angina, coronary/peripheral artery bypass graft, or cerebrovascular accident.
* Patients with New York Heart Association Class III or IV heart failure.
* Inability to comply with protocol mandated hospitalizations and restrictions
* Patients who are pregnant, breast-feeding, or intending to become pregnant during the study.
* Prior solid organ or allogeneic stem cell transplantation
* History of known or suspected hemophagocytic lymphohistiocytosis (HLH).
* History of autoimmune disease, including but not limited to myocarditis, pneumonitis, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis • Patients with a remote history of, or well controlled, autoimmune disease may be eligible to enroll after consultation with the study PI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2023-07-18 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
End of Treatment (EOT) Complete Metabolic Response (CMR) Rate | (Cycle 1 = 36 days, cycle 2 - 12 = 21 days), up to 267 days
  EOT CMR rate defined as the proportion of participants achieving CR per PET/CT Lugano 2014 criteria (protocol appendix B) at the EOT assessment: PET-CT, score 1, 2, or 3 with or without a residual mass on a 5-point scale (5PS).

SECONDARY OUTCOMES:
Best Partial Metabolic Response (PMR) Rate | (Cycle 1 = 36 days, cycle 2 - 12 = 21 days), up to 267 days
  Best PMR rate defined as the proportion of participants achieving PR per Lugano 2014 criteria (protocol appendix B) ever on treatment: PET-CT Score 4 or 5 with reduced uptake compared with baseline and residual mass(es) of any size or on CT, ≥ 50% decrease in SPD of up to 6 target measurable nodes and extranodal sites; no increase in non-measured lesions; spleen if enlarged must have regressed by >50% in length beyond normal.
Best Complete Metabolic Response (CMR) Rate | (Cycle 1 = 36 days, cycle 2 - 12 = 21 days), up to 267 days
  Best CMR rate defined as the proportion of participants achieving CR per Lugano 2014 criteria (protocol appendix B) ever on treatment.
Best Objective Metabolic Response (OMR) Rate | (Cycle 1 = 36 days, cycle 2 - 12 = 21 days), up to 267 days
  Best OMR rate defined as the proportion of participants achieving CR or partial response (PR) per Lugano 2014 criteria (protocol appendix B) ever on treatment.
EOT Partial Metabolic Response (PMR) Rate | (Cycle 1 = 36 days, cycle 2 - 12 = 21 days), up to 267 days
  EOT PMR rate defined as the proportion of participants achieving PR per PET/CT Lugano 2014 criteria (protocol appendix B) at the EOT assessment: PET-CT Score 4 or 5 with reduced uptake compared with baseline and residual mass(es).
EOT Objective Metabolic Response (OMR) Rate | (Cycle 1 = 36 days, cycle 2 - 12 = 21 days), up to 267 days
  EOT OMR rate defined as the proportion of participants achieving CR or partial response (PR) per PET/CT Lugano 2014 criteria (protocol appendix B) at the EOT assessment.
2-year Duration of Response (DOR) | 2 years
  2-year DOR is a probability estimated using the Kaplan Meier method; DOR is defined as the time measurement criteria are met for CR or PR (whichever is first recorded) per Lugano 2014 criteria (protocol Appendix B) until the first date that recurrent or progressive disease is objectively documented, or death due to any cause. CR and PR participants without events reported are censored at the last disease evaluation.
2-year Duration of Complete Response (DOCR) | 2 years
  2-year DOCR is a probability estimated using the Kaplan Meier method; DOCR is defined as the time measurement criteria are met for CR per Lugano 2014 criteria (protocol Appendix B) until the first date that recurrent or progressive disease is objectively documented, or death due to any cause. CR participants without events reported are censored at the last disease evaluation.
2-year Progression-free Survival (PFS) | 2 years
  2-year PFS is a probability estimated using the Kaplan Meier method; PFS is defined as the duration of time from study entry to documented disease progression (PD) or death. PD defined by Lugano 2014 criteria (protocol Appendix B).
2-year Time-to-Next Treatment (TTNT) | 2 years
  2-y TTNT is a probability estimated using the Kaplan Meier method; TTNT is defined as the duration of time from the first dose of treatment until the time of initiation of new therapy, or censored at the date of last contact.
2-year Overall Survival (OS) | 2 years
  2-year OS is a probability estimated using the Kaplan-Meier method; OS is defined as the time from study entry to death, or censored at date last known alive.
Incidence of Histological Transformation | up to 10 years
  Histological transformation was defined as participants who have a biopsy showing diffuse large B-cell lymphoma (DLBCL). Incidence is the number of participants with histological transformation during or after treatment.
Number of Participants with Cytokine Release Syndrome (CRS) by Grade | (Cycle 1 = 36 days, cycle 2 - 12 = 21 days), up to 267 days + 30 days
  All grade CRS AEs regardless of attribution based on American Society of Transplantation and Cellular Therapy [ASTCT] Consensus grading as reported on case report forms are counted and maximum grade tabulated. Incidence by grade is then tabulated as the number of participants ever experiencing maximum grade during the time of observation.
Grade 3-5 Treatment-Related CRS Rate | (Cycle 1 = 36 days, cycle 2 - 12 = 21 days), up to 267 days + 30 days
  All grade 3-5 CRS AEs with attribution of probably, possibly or definitely-related to treatment based on American Society of Transplantation and Cellular Therapy [ASTCT] Consensus grading as reported on case report forms were counted. Rate is the proportion of treated participants experiencing at least one treatment-related grade 3-5 CRS AE of any type during the time of observation.
Number of Participants with Neurotoxicity by Grade | (Cycle 1 = 36 days, cycle 2 - 12 = 21 days), up to 267 days + 30 days
  All grade neurotoxicity AEs regardless of attribution based on CTCAEv5 as reported on case report forms are counted and maximum grade tabulated. Incidence by grade is then tabulated as the number of participants ever experiencing maximum grade during the time of observation.
Grade 3-5 Treatment-Related Neurotoxicity Rate | (Cycle 1 = 36 days, cycle 2 - 12 = 21 days), up to 267 days + 30 days
  All grade 3-5 neurotoxicity AEs with attribution of probably, possibly or definitely-related to treatment based on CTCAEv5 as reported on case report forms were counted. Rate is the proportion of treated participants experiencing at least one treatment-related grade 3-5 neurotoxicity AE of any type during the time of observation.
Grade 3-5 Toxicity Rate | (Cycle 1 = 36 days, cycle 2 - 12 = 21 days), up to 267 days + 30 days
  All grade 3-5 AEs regardless of attribution based on CTCAEv5 as reported on case report forms were counted. Rate is the proportion of treated participants experiencing at least one grade 3-5 AE of any type during the time of observation.
Grade 3-5 Treatment-Related Toxicity Rate | (Cycle 1 = 36 days, cycle 2 - 12 = 21 days), up to 267 days + 30 days
  All grade 3-5 AEs with attribution of probably, possibly or definitely-related to treatment based on CTCAEv5 as reported on case report forms were counted. Rate is the proportion of treated participants experiencing at least one treatment-related grade 3-5 AE of any type during the time of observation.
Grade 2-5 Treatment-Related Toxicity Rate | (Cycle 1 = 36 days, cycle 2 - 12 = 21 days), up to 267 days + 30 days
  All grade 2-5 AEs with attribution of probably, possibly or definitely-related to treatment based on CTCAEv5 as reported on case report forms were counted. Rate is the proportion of treated participants experiencing at least one treatment-related grade 2-5 AE of any type during the time of observation.

CONTACTS AND LOCATIONS:
Overall Officials: Reid Merryman, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (4):
- United States (4):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Columbia University Irving Medical Center, New York, New York
  - Mount Sinai Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu